CLINICAL TRIAL: NCT01955759
Title: Pharmacologic Prophylaxis for Atrial Fibrillation Following Coronary By-Pass Surgery
Brief Title: Atrial Fibrillation and By-pass Surgery
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Heart Center BH Tuzla (Other)
Responsible Party: Principal Investigator, Enes Osmanović, Mr.med.sc.Dr Enes Osmanovic, Heart Center BH Tuzla
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 0115/09 - (2013)
Record Dates: First submitted 2013-09-21; First posted 2013-10-07 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Patients With Coronary Artery Disease Scheduled for by Pass Surgery
MeSH Terms: interventions — Amiodarone; Rosuvastatin Calcium; Bisoprolol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- beta blocker and amiodarone (Experimental): The inteventin will be that patients will receive beta blocker Bisoprolol in adjusted dose + Amiodarone per os starting 7 days before coronary by-pass surgery, 200 mg. x 3 tab, followed by 200 mg x 2 tab per os starting on the second postoperative day untill discharge
  Interventions: Drug: Amiodarone tab 200 mg x 3; Drug: beta blockers Bisoprolol in adjusted dose
- beta blocker and statin (Experimental): The intervention will be that patients will receive beta blocker (Bisoprolol tab in adjusted dose)+ Rosuvastatin 20 mg. x 1 starting 7 days before coronary by-pass surgry untill discharge.
  Interventions: Drug: rosuvastatin 20 mg tab x1; Drug: beta blockers Bisoprolol in adjusted dose
- beta blocker (Placebo Comparator): Patients will receive beta blocker (Bisoprolol tab in adjusted dose).
  Interventions: Drug: beta blockers Bisoprolol in adjusted dose

INTERVENTIONS:
Drug: Amiodarone tab 200 mg x 3 — starting 7 days before coronary by-pass surgery per os 200 mg. x 3 tab, followed by 200 mg x 2 tab per os starting on the second postoperative day untill discharge
  Other Names: cordarone
  Arms: beta blocker and amiodarone
Drug: rosuvastatin 20 mg tab x1 — starting 7 days before coronary by-pass surgery
  Other Names: crestor
  Arms: beta blocker and statin
Drug: beta blockers Bisoprolol in adjusted dose — starting 7 days befoe coronary by-pass surgery
  Other Names: zebeta

SUMMARY:
The aim of the study is to evaluate whether combined therapy with beta-blocker, amiodarone and statine is better than beta-blocker alone for the prevention of atrial fibrillation after coronary by-pass surgery.

ELIGIBILITY:
Inclusion Criteria:

* significant coronary disease, sinus rhythm

Exclusion Criteria:

* valvular disease, former by-pass surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-12 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
atrial fibrillation | 10 days on average during hospital stay after coronary by-pass surgery
  outcome will be number of patients free from atrial fibrillation.

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Center BH, Tuzla, TK, Bosnia and Herzegovina